CLINICAL TRIAL: NCT01571310
Title: Effect of Breakfast Omission on Postprandial Glycemia After Lunch and Dinner in T2D
Brief Title: Effect of Breakfast or Omission of Breakfast in T2D
Acronym: OB-B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel Aviv University (Other)
Collaborators: Hospital de Clinicas Caracas (Other)
Responsible Party: Principal Investigator, Daniela Jakubowicz, Prof. Daniela Jakubowicz MD, Tel Aviv University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: HCCCBI 017-2007-112
Record Dates: First submitted 2012-03-30; First posted 2012-04-05 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Breakfast

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Omitted Breakfast (Experimental): Experimental: The patients in Omitted Breakfast day will omit the breakfast and will continue the fast until noon. Thereafter will eat Lunch at 13;30 and Dinner at 19:00
  Interventions: Other: Omitted Breakfast; Other: Breakfast
- Breakfast (Active Comparator): The patients in Breakfast day will consume breakfast at 8:00 and then lunch at 13;30 and dinner at 19:00
  Interventions: Other: Omitted Breakfast; Other: Breakfast

INTERVENTIONS:
Other: Omitted Breakfast — Experimental:The patients in Omitted Breakfast day will omit the breakfast and will continue the overnight fast until lunch. They will eat only lunch (700 kcal) at 13:30 and dinner (700 kcal) at 19:00
  Other Names: Omission of Breakfast
Other: Breakfast — In the Active Comparator: The patients in the Breakfast day will consume breakfast (700 kcal) at 8:00 , lunch (700 kcal) at 13:30 and dinner (700 kcal) at 19:00
  (YesB): The patients in YesB will eat all three mealswill consume three meals:
  Other Names: Breakfast consupmtion

SUMMARY:
The investigators will explore the effect of omission of breakfast on postprandial hyperglycemia and insulin and intact GLP-1 response after subsequent meals in type 2 diabetic patients

DETAILED DESCRIPTION:
In obesity and in type 2 diabetes eating behavior especially the lack of breakfast promote weight gain, increase hunger and carbohydrate craving.

The present study is designed to address whether in T2D, a change in meal timing; specifically, by adding calories, protein and carbohydrates to the breakfast vs.the omission of breakfast will influence the postprandial elevation of glucose, insulin, intact GLP-1, glucagon and free fatty acids (FFA) after subsequent meals at lunch and dinner.

The investigators expect that compared to the day with breakfast condition the day when the breakfast will be omitted the postprandial glucose , free fattly acids, and glucagon response after lunch and dinner will be significative higher while insulin and intact GLP-1 response after lunch and dinner will be reduced

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetics for < 10yr
2. HbA1C: 7-9 %
3. BMI: 22 to 35 kg/m2)
4. Age: ≥30 and ≤70 years of age
5. Habitually eat breakfast
6. Naïve or treated with oral antidiabetic drugs and those with anti-hypertensive and lipid-lowering medication
7. Those treated with insulin or GLP-1 analogs or having major liver, heart or kidney illnesses will be excluded.
8. Usually wake up between 06:00 and 07:00 and go to sleep between 22:00 and 24:00.
9. Not dieting and no change in body weight >10 lb = 4.5 kg within the last 6 months
10. Stable physical activity pattern during the three months immediately preceding study initiation
11. Normal liver and kidney function 12 No metabolic disease other then diabetes

13. Usually wakes up between 05:00 and 07:00 and goes to sleep between 22:00 and 24:00.

15. Normal TSH and FT4 levels 16. Acceptable health based on interview, medical history, physical examination, and laboratory tests 17. Those who provide signed informed consent

Exclusion Criteria:

1. Type 1 diabetes
2. Pulmonary disease, psychiatric, immunological, neoplastic diseases or severe diabetic complications, such as cardiovascular disease, cerebrovascular disease, proliferative diabetic retinopathy, gastroparesis or underwent bariatric surgery.
3. Abnormal liver function tests defined as an increase by a factor of at least 2 above the upper normal limit of alanine aminotransferase and/or aspartate
4. Anemia (Hg > 10g/dL)
5. Serum creatinine level > 1.5 mg/dl
6. Pregnant or lactating
7. Participating in another dietary program or use of weight-loss medications
8. Documented or suspected history (within one year) of illicit drug abuse or alcoholism.
9. Use of psychotropic or anoretic medication during the month immediately prior to study onset

13.Work shifts within the last 5 years and did not cross time zones within the last month of the study.

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Postprandial Glucose Response | 12 weeks
  Postprandial Glucose response will be measure after lunch and dinner

SECONDARY OUTCOMES:
Postprandial Insulin Response | 12 weeks
  Postprandial Insulin response will be measure after lunch and dinner
Postprandial intact-GLP-1 Response | 12 weeks
  Postprandial intact-GLP-1 response will be measure after lunch and dinner
Postprandial Glucagon Response | 12 weeks
  Postprandial Glucagon response will be measure after lunch and dinner
Postprandial Free Fatty Acids Response | 12 weeks
  Postprandial Free Fatty Acids response will be measure after lunch and dinner

CONTACTS AND LOCATIONS:
Overall Officials: Julio Wainstein, MD, Principal Investigator — Head of Diabetes Unit E. Wolfson Medical Center Israel; Daniela Jakubowicz, MD, Principal Investigator — Hospital de Clinicas Caracas, Venezuela
Locations (2):
- Daniela Jakubowicz, Holon, N/A = Not Applicable, Israel
- Daniela Jakubowicz, Caracas, Venezuela

REFERENCES:
- [Derived] Allaf M, Elghazaly H, Mohamed OG, Fareen MFK, Zaman S, Salmasi AM, Tsilidis K, Dehghan A. Intermittent fasting for the prevention of cardiovascular disease. Cochrane Database Syst Rev. 2021 Jan 29;1(1):CD013496. doi: 10.1002/14651858.CD013496.pub2. PMID 33512717